CLINICAL TRIAL: NCT01151488
Title: Impact of Nutrition and Exercise on Glucose Metabolism, Inflammation, and Body Composition in Older Breast Cancer Survivors
Brief Title: Nutrition, Exercise, and Breast Cancer Survivorship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Alice S. Ryan, PhD, Professor, Baltimore VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00045555; P30AG028747 (NIH)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer Survivorship; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistance Training (Experimental): 16 weeks of moderate intensity resistance training, 3x/week
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Resistance Training — RT 3x/wk for 4 months
  Other Names: Exercise

SUMMARY:
The purpose of the study is to examine the effects of resistance training on the reasons (mechanisms) underlying the development of fatigue, muscle weakness and wasting (sarcopenia), and impaired physical functioning (poor balance and walking) associated with breast cancer survivorship.

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed cancer in women, representing 26% of all female cancers. It is also the second leading cause of cancer related deaths in the US for women. Side effects of the cancer and treatment therapies may result in inactivity and inadequate intakes of various nutrients, including protein and vitamin D, associated with cardiovascular disease (CVD) and type 2 diabetes. High concentrations of systemic and local inflammation correlate well with CVD and diabetes risk. There is substantial evidence to support that incorporating physical activity and nutrition into one's lifestyle can reduce inflammation and, ultimately, the progression to CVD and diabetes. Understanding the role of exercise and diet management in the health of breast cancer survivors will allow us to translate these findings into therapy guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of previous breast cancer
* Three months post active cancer therapy (i.e. radiation/chemotherapy)
* Non smoker (non smoking for at least 12 months: cigarettes, cigars, pipes)
* 45-80 years of age
* Menopause over one year (absence of menses for 12 months or greater)
* Sedentary lifestyle (structured physical activity </= 2x per week)
* BMI >/=18 and <50 kg/m2

Exclusion Criteria:

* Unstable lymphedema (no intensive therapy, no recorded 10% change in arm volume or circumference, no more than one lymphedema-related infection requiring antibiotics and no change in ADLs due to a lymphedema exacerbation for the past 3 months)
* Plans for surgery (e.g., breast reconstruction) during the study period
* Evidence of recurrent cancer or metastases
* Symptomatic heart disease, CAD, CHF, or uncontrolled hypertension (SBP over 180 mm HG) unless medically stabilized
* Abnormal renal function (BUN above 40 mg/dl, Cr above 1.3 mg/dl, CrCl<60mg/dl)
* Anemia HCT below 30 mg/dl, platelets below 100,000/cm3
* History of seizures or taking anti-seizure or anti convulsion medication
* Untreated dyslipidemia with National Cholesterol ATPIII 10 year cardiac risk score greater than 10% (www.nhlbi.nih.gov/guidelines/cholesterol/atp3upd04.htm)
* Allergic to lidocaine
* Abnormal liver function
* Abnormal response to exercise test (ST segment depression greater than 2mm, chest pain, significant arrhythmias, extreme shortness of breath, cyanosis, exercising BP above 240/120 mm HG, or other contraindications to exercise) confirmed with further diagnostic evaluations.
* Type 1 diabetes; insulin treatment for diabetes, poorly controlled diabetes, HgA1c>10%
* Taking oral steroids, warfarin, or other medications interfering with fat/muscle metabolism that may not be safely discontinued temporarily for specific procedures (i.e. for 72 hours prior)
* MMSE below 24, dementia, or unstable clinical depression by exam
* Chronic pulmonary disease (on supplemental O2)
* Metal implants or devices (i.e. pacemaker) if undergoing CT scan
* Participant is, in the opinion of the investigator, unable to adhere to the study protocol due to medical or orthopedic conditions that limit ability to exercise or travel to the Baltimore VA for protocol procedures
* Aerobically trained with VO2max greater than 2 SD above age-adjusted mean
* Alcohol consumption greater than 3 oz. liquor, 3x4 oz glass of wine, or 2x12 oz beers per day, by self report

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
muscle performance | change in muscle area between baseline and 16 weeks
  muscle strength

SECONDARY OUTCOMES:
glucose tolerance | change in glucose levels between baseline and 16 weeks
  glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P Goldberg, M.D., Principal Investigator — Baltimore VAMC/GRECC
Locations (1):
- Baltimore VAMC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No